CLINICAL TRIAL: NCT06714734
Title: Thromboembolic and Hemorrhagic Complications of Anticoagulant Treatment in Patients With CAT (Cancer Associated Thrombosis)
Brief Title: Thromboembolic and Hemorrhagic Complications of Anticoagulant Treatment in Patients With CAT
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: CAT-Ther
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Venous Thromboembolism
Keywords: TVP; CAT
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is classified as an observational pharmacological study, spontaneous, monocentric, and both retrospective and prospective for adult patients with a diagnosis of venous thromboembolism in the context of neoplasia, followed at the SSD Angiology and Coagulation Disorders of the IRCCS Azienda Ospedaliero-Universitaria di Bologna and The Cardiovascular Medicine Department, specifically the Angiology Unit, of the IRCCS Arcispedale S. Maria Nuova in Reggio Emilia, from 01/01/2016 to 30/06/2027. The study, including data analysis, is expected to conclude by 31/12/2027.

Patients were treated according to clinical practice, in accordance with the physician's judgment and the information provided in the product's technical datasheet for any concomitant therapies administered as per clinical practice.

The primary objective of the study is to evaluate the frequency of thrombotic and hemorrhagic complications during treatment with low molecular weight heparin or direct oral anticoagulants in patients with venous thromboembolism and solid and hematological neoplasms attending outpatient care at the SSD Angiology and Coagulation Disorders of the IRCCS AOUBO and The Cardiovascular Medicine Department, specifically the Angiology Unit, of the IRCCS Arcispedale S. Maria Nuova in Reggio Emilia, following the initiation of anticoagulant therapy (LMWH or DOACs).

The secondary objectives of the study are:

* To identify risk factors for hemorrhagic complications and bleeding risk during anticoagulant treatment for CAT;
* To assess the applicability and reliability of a score, which is not currently in use in clinical practice, without impacting the care process and clinical decisions, in a prospective cohort of patients with CAT.

DETAILED DESCRIPTION:
The study is classified as an observational study involving the use of medication, spontaneous, multicentric, retrospective, and prospective for adult patients with a diagnosis of venous thromboembolism in the context of neoplasia, followed at the SSD Angiology and Coagulation Disorders of the IRCCS Azienda Ospedaliero-Universitaria di Bologna and The Cardiovascular Medicine Department, specifically the Angiology Unit, of the IRCCS Arcispedale S. Maria Nuova in Reggio Emilia.

The study, including data analysis, is expected to conclude by 31/12/2027. Patients have been and will be treated according to clinical practice, in accordance with the physician's judgment and the information provided in the technical datasheet of each product used for any concomitant therapies administered as per clinical practice. The diagnostic-therapeutic pathway for patients will not be influenced in any way by the results of the tissue tests performed for the purposes of the study.

Additionally, patients have been and will be followed according to the usual schedule defined by current clinical practice and will undergo all standard diagnostic investigations, both invasive and non-invasive, as prescribed by current clinical practice.

All adult patients with a diagnosis of venous thromboembolism in the context of neoplasia, followed at the SSD Angiology and Coagulation Disorders of the IRCCS Azienda Ospedaliero-Universitaria di Bologna and The Cardiovascular Medicine Department, specifically the Angiology Unit, of the IRCCS Arcispedale S. Maria Nuova in Reggio Emilia, will be enrolled from 01/01/2016 to 30/06/2027.

Each patient will be followed according to standard clinical-care practice, with a follow-up of at least 6 months considered for the purposes of the study.

Considering that the monthly attendance of patients at the Consultation Clinic of the SSD Angiology and Coagulation Disorders of the IRCCS AOUBO and The Cardiovascular Medicine Department, specifically the Angiology Unit, of the IRCCS Arcispedale S. Maria Nuova in Reggio Emilia is approximately 50 patients, based on the inclusion/exclusion criteria, it is estimated that about 1,000 patients with a diagnosis of VTE in the context of neoplasia can be enrolled.

This sample size is considered sufficient to achieve the primary objective of the study.

The primary objective is to evaluate the frequency of thrombotic and hemorrhagic complications during treatment with low molecular weight heparin or direct oral anticoagulants in patients with venous thromboembolism and solid and hematological neoplasms, followed in outpatient care at the SSD Angiology and Coagulation Disorders of the IRCCS AOUBO and The Cardiovascular Medicine Department, specifically the Angiology Unit, of the IRCCS Arcispedale S. Maria Nuova in Reggio Emilia, following the initiation of anticoagulant therapy (LMWH or DOACs).

The secondary objectives are:

* To identify risk factors for hemorrhagic complications and bleeding risk during anticoagulant treatment for CAT,
* To assess the applicability and reliability of a score, which is not currently used in clinical practice, without affecting the care process and clinical decisions, in a prospective cohort of patients with CAT.

The data available in the literature concern the use of anticoagulants (LMWH or DOACs) in patients with a confirmed diagnosis of venous thromboembolism in the context of neoplasia. However, it is necessary to stratify these patients in order to identify those who are more or less at risk of complications, in order to provide a more targeted therapeutic approach.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of venous thrombosis at any site
* Diagnosis of CVC-related venous thrombosis
* Diagnosis of pulmonary embolism, both symptomatic and incidental
* Diagnosis of solid or hematological neoplasm, either under treatment or active
* Obtaining of Informed Consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with a diagnosis of venous thromboembolism in the context of neoplasia, followed at the SSD Angiology and Coagulation Disorders of the IRCCS Azienda Ospedaliero-Universitaria di Bologna and The Cardiovascular Medicine Department, specifically the Angiology Unit, of the IRCCS Arcispedale S. Maria Nuova in Reggio Emilia, will be enrolled from 01/01/2016 to 30/06/2027. Each patient will be followed according to standard clinical-care practice, with a follow-up of at least 6 months considered for the purposes of the study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-01-02 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Thrombotic and Hemorrhagic Complications During Treatment with Low Molecular Weight Heparin or Direct Oral Anticoagulants in Patients with Venous Thromboembolism and Neoplasms | From enrollment to the end of treatment at 6 months
  To evaluate the frequency of thrombotic and hemorrhagic complications during treatment with low molecular weight heparin or direct oral anticoagulants in patients with venous thromboembolism and solid and hematological neoplasms, followed in outpatient care at the SSD Angiology and Coagulation Disorders of the IRCCS AOUBO and The Cardiovascular Medicine Department, specifically the Angiology Unit, of the IRCCS Arcispedale S. Maria Nuova in Reggio Emilia, following the initiation of anticoagulant therapy (LMWH or DOACs).

SECONDARY OUTCOMES:
Risk factors for hemorrhagic complications and bleeding risk | From enrollment to the end of treatment at 6 months
  To identify risk factors for hemorrhagic complications and bleeding risk during anticoagulant treatment for CAT.
Applicability and reliability of a score | From enrollment to the end of treatment at 6 months
  To assess the applicability and reliability of a score, which is not currently used in clinical practice, without impacting the care process and clinical decisions, in a prospective cohort of patients with CAT.

CONTACTS AND LOCATIONS:
Overall Officials: Benilde Cosmi, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (2):
- Italy (2):
  - IRCCS Azianda Ospedaliero-Universitaria di Bologna, Bologna
  - IRCCS Arcispedale S. Maria Nuova di Reggio Emilia, Reggio Emilia